CLINICAL TRIAL: NCT00772954
Title: A Phase I Randomized, Placebo-Controlled, Double-Blind, Dose Ranging Study of the Safety, Tolerability and Immunogenicity of Two Doses of a Clostridium Difficile Toxoid Vaccine, Alum Adsorbed, in Healthy Adult Volunteers (18 - 55 Years)
Brief Title: Phase I Randomized, Placebo-Controlled, Double-Blind, Dose Ranging Study, Safety, Tolerability and Immunogenicity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Issues with CTM stability.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-030-010
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-04

CONDITIONS: Clostridium Difficile Infection; Clostridium Difficile Diarrhea
Keywords: Clostridium difficile diarrhea; Clostridium difficile toxoid vaccine
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo vaccine group (Placebo Comparator): Participants scheduled to receive a dose of placebo vaccine on Day 0, Day 28, and Day 56, respectively.
  Interventions: Biological: Vaccine diluent buffer
- Clostridium Difficile Vaccine Group 1 (Experimental): Participants scheduled to receive a dose of 50 μg Clostridium Difficile vaccine on Day 0, Day 28, and Day 56, respectively.
  Interventions: Biological: Clostridium difficile toxoid vaccine (50 μg)
- Clostridium Difficile Vaccine Group 2 (Experimental): Participants scheduled to receive a dose of 100 μg Clostridium Difficile vaccine on Day 0, Day 28, and Day 56, respectively.
  Interventions: Biological: Clostridium difficile toxoid vaccine (100 μg)

INTERVENTIONS:
Biological: Vaccine diluent buffer — 0.5 mL, Intramuscular at Day 0, Day 28 and Day 56, respectively.
  Arms: Placebo vaccine group
Biological: Clostridium difficile toxoid vaccine (50 μg) — 0.5 mL, Intramuscular at Day 0, Day 28 and Day 56, respectively.
  Arms: Clostridium Difficile Vaccine Group 1
Biological: Clostridium difficile toxoid vaccine (100 μg) — 0.5 mL, Intramuscular on Day 0, Day 28 and Day 56, respectively.
  Arms: Clostridium Difficile Vaccine Group 2

SUMMARY:
This Phase I, randomized, placebo-controlled, double-blinded, dose ranging study to assess the safety, tolerability, and immunogenicity of 2 dose levels of C. difficile vaccine. Population: healthy male and female adults, 18 to 55 years old.

DETAILED DESCRIPTION:
This was a Phase I, randomized, placebo-controlled, double-blinded, dose ranging study designed to assess the safety, tolerability, and immunogenicity of C. difficile vaccine. The study was conducted in healthy male and female adults, 18 to 55 years old. Subjects was randomly assigned on Day 0 to receive one of two doses of C. difficile vaccine (50 or 100 mcg) or placebo (vehicle control containing alum).

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females, 18 - 55 years in good general health

Exclusion Criteria:

* Evidence of current C. difficile infection, as determined by a positive stool C. difficile cytotoxin assay at screening
* Evidence of any previous antibiotic-associated diarrhea caused by any etiology including C. difficile that required medical intervention or medication
* Active or inactive irritable bowel disease, chronic abdominal pain, chronic diarrhea of any etiology, or inflammatory bowel disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis N Morrison, D.O., Principal Investigator — Bio-Kinetic Clinical Applications, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled on 28 March 2006 in 2 clinical centers in the US.
Pre-assignment Details: A total of 36 participants who met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- Placebo Vaccine Group: Participants received a dose of placebo (vaccine diluent) on Day 0 and Day 28.
- Clostridium Difficile Toxoid Vaccine Group 1: Participants received a dose of 50 μg Clostridium difficile toxoid vaccine on Day 0 and Day 28.
- Clostridium Difficile Toxoid Vaccine Group 2: Participants received a dose of 100 μg Clostridium difficile toxoid vaccine on Day 0 and Day 28.
Period: Overall Study
Arm/Group | Placebo Vaccine Group | Clostridium Difficile Toxoid Vaccine Group 1 | Clostridium Difficile Toxoid Vaccine Group 2
Started | 12 | 12 | 12
Completed | 12 | 12 | 11
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Vaccine Group | Clostridium Difficile Toxoid Vaccine Group 1 | Clostridium Difficile Toxoid Vaccine Group 2 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (12.98) | 36.9 (12.67) | 30.0 (8.57) | 35.1 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 5 | 23
  Male | 5 | 1 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events Post-vaccination With One of Two Formulations of Clostridium Difficile Toxoid Vaccine or a Placebo Vaccine.
Time Frame: Day 0 up to 70 days post first vaccination
Population: Safety assessments were on the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo Vaccine Group | Clostridium Difficile Toxoid Vaccine Group 1 | Clostridium Difficile Toxoid Vaccine Group 2
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Injection site pain | 7 | 12 | 9
  Headache | 5 | 4 | 5
  Blood potassium decreased | 1 | 4 | 3
  Protein urine present | 1 | 4 | 3
  White blood cell count increased | 1 | 4 | 3
  Diarrhoea | 3 | 3 | 2
  Fatigue | 3 | 3 | 2
  Myalgia | 1 | 5 | 1
  White blood cells urine positive | 2 | 2 | 3
  Eosinophil count increased | 3 | 1 | 3
  Abdominal pain | 2 | 1 | 3
  Injection site erythema | 2 | 3 | 1
  Red blood cells urine positive | 2 | 2 | 2
  Injection site swelling | 0 | 4 | 1
  Injection site warmth | 0 | 2 | 2
  Malaise | 0 | 3 | 0
  Blood urea increased | 2 | 1 | 0
  Sinus congestion | 2 | 0 | 1
  Urine ketone body present | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination 1 (Day 0) to up to 8 months post-vaccination.
Arm/Group | Placebo Vaccine Group | Clostridium Difficile Toxoid Vaccine Group 1 | Clostridium Difficile Toxoid Vaccine Group 2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 12/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Vaccine Group (N=12) | Clostridium Difficile Toxoid Vaccine Group 1 (N=12) | Clostridium Difficile Toxoid Vaccine Group 2 (N=12)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3
Injection site pain (General disorders) | 7 | 12 | 9
Fatigue (General disorders) | 3 | 3 | 2
Injection site erythema (General disorders) | 2 | 3 | 1
Injection site swelling (General disorders) | 0 | 4 | 1
Injection site warmth (General disorders) | 0 | 2 | 2
Malaise (General disorders) | 0 | 3 | 0
Blood potassium decreased (Investigations) | 1 | 4 | 3
Protein urine present (Investigations) | 1 | 4 | 3
White blood cell count increased (Investigations) | 1 | 4 | 3
White blood cells urine positive (Investigations) | 2 | 2 | 3
Eosinophil count increased (Investigations) | 3 | 1 | 3
Red blood cells urine positive (Investigations) | 2 | 2 | 2
Blood urea increased (Investigations) | 2 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Headache (Nervous system disorders) | 5 | 4 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Injection site hemorrhage (General disorders) | 0 | 1 | 0
Injection site induration (General disorders) | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 1
Monocyte count increased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early in light of issues with CTM stability. All other study procedures and visits were performed per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications